CLINICAL TRIAL: NCT01656174
Title: Procleix® Dengue Virus Assay Testing of Individual Donor Samples From Puerto Rican Blood Donors - American Red Cross
Status: Completed | Type: Observational
Sponsor: Gen-Probe, Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: DENVTS-US12-001
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment
  Interventions: Device: Procleix Dengue Virus Assay

INTERVENTIONS:
Device: Procleix Dengue Virus Assay — in vitro diagnostic assay

SUMMARY:
The objective of this study is to test individual donor samples (IDSs) with the investigational Dengue Assay on the TIGRIS System and to further characterize the Dengue Assay in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Donor must meet all the blood collection sites' standard eligibility requirements.
* Donor and/or legally authorized representative must be willing to undergo the site's routine informed consent process prior to study participation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: volunteer blood donors from Puerto Rico
Sampling Method: Non-Probability Sample
Enrollment: 35035 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Qualitative detection of ribosomal RNA from Dengue Virus in plasma specimens from individual human donors, including volunteer donors of whole blood and blood components, and other living donors. | Approximately three years

CONTACTS AND LOCATIONS:
Overall Officials: Renee Wait, Study Director — Gen-Probe, Incorporated
Locations (2):
- United States (2):
  - Creative Testing Solutions, Tempe, Arizona
  - American Red Cross National Testing Laboratory, Charlotte, North Carolina